CLINICAL TRIAL: NCT01874561
Title: A Single-Center, Double-Blind, Randomized, Placebo- and Positive-Controlled, Parallel Group, Thorough QT/QTc Study to Evaluate the Effect of Custirsen (640 mg) on Cardiac Repolarization in Healthy Men
Brief Title: Thorough QT/QTc (Corrected QT Interval) Study to Evaluate the Effect of Custirsen on Cardiac Repolarization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV1011-TQT-108
Record Dates: First submitted 2013-05-01; First posted 2013-06-11 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Cardiac Conduction and Repolarization
Keywords: Custirsen sodium; TV1011; OGX-011; Thorough QT study; cancer
MeSH Terms: conditions — Neoplasms | interventions — OGX-011; Saline Solution; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Group 1: investigational product (custirsen) will receive:
  * 320 mg of custirsen + 5 mg of dexamethasone on day 1
  * 480 mg of custirsen + 5 mg of dexamethasone on day 3
  * 640 mg of custirsen + 3 mg of dexamethasone on day 5
  * 640 mg of custirsen on day 7 under fasting conditions
  Interventions: Drug: Custirsen
- Group 2 (Placebo Comparator): Group 2: placebo (normal saline) will receive:
  * placebo + 5 mg of dexamethasone on day 1
  * placebo + 5 mg of dexamethasone on day 3
  * placebo + 3 mg of dexamethasone on day 5
  * placebo on day 7 under fasting conditions
  Interventions: Drug: Placebo
- Group 3 (Active Comparator): Group 3: positive control (moxifloxacin) will receive:
  * placebo + 5 mg of dexamethasone on day 1
  * placebo + 5 mg of dexamethasone on day 3
  * placebo + 3 mg of dexamethasone on day 5
  * 400 mg of moxifloxacin + placebo (immediately after moxifloxacin administration) on day 7 under fasting conditions
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Custirsen — Custirsen will be administered iv using an infusion pump over a 2-hour period.
  Other Names: custirsen sodium
  Arms: Group 1
Drug: Placebo — Placebo (commercially available normal saline) will be administered iv using an infusion pump over a 2-hour period.
  Other Names: Normal saline
  Arms: Group 2
Drug: Moxifloxacin — Moxifloxacin (400 mg) will be administered orally with 240 mL of room temperature still water.
  Arms: Group 3

SUMMARY:
This is a 3-arm, parallel-group, active- and placebo-controlled, double-blind, randomized study, to compare treatment with intravenous custirsen at 640 mg (highest intended therapeutic dose) with placebo. The purpose of this study is to assess the effect of custirsen treatment on cardiac conduction and repolarization (electrical activity of the heart) in healthy subjects. The positive control employed to demonstrate assay sensitivity consists of a group receiving a single oral dose of 400 mg moxifloxacin on day 7. The moxifloxacin arm is un-blinded but the ECG readings are blinded.

DETAILED DESCRIPTION:
The effects of custirsen will be evaluated following administration of a single dose following dose-titration period combined with dexamethasone pretreatment. On days -1 and 7, subjects will undergo a full ECG assessment for 24 hours. On day 1, randomization and assignment to the treatment groups will be performed prior to drug administration. Subjects will remain in the study center throughout the treatment period. All subjects will be discharged at the end of day 8 procedures, 24 hours after the last dose of custirsen has been administered. Subjects in groups 1 and 2 will return for an additional visit on day 9, 10 and 14 (±2 days) (approximately 7 days after the last study drug administration). Subjects in group 3 will not return for a follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a man aged 18 through 45 years of age with a body mass index (BMI) of 18 through 30 kg/m2 at screening.
2. The subject is in good health as determined by medical history, ECG, vital signs measurements, physical examination, and clinical laboratory tests.
3. The subject must be able to understand and comply with the requirements of the study (eg, all medication, dietary, exercise, tobacco, and alcohol restrictions).
4. The subject must provide written informed consent to participate in the study after reading the information and consent form, and after having an opportunity to discuss the study with the investigator or delegate.
5. Other inclusion criteria apply.

Exclusion Criteria:

1. Exclusion criteria related to ECG findings include the following:

   * The subject has an ECG abnormality that may interfere with the accurate assessment of the QT interval, including intraventricular conduction delays (QRS >120 msec or PR >200 as measured at the screening and check-in visits) and complete or incomplete bundle branch blocks.
   * The subject has a resting QTcF interval of ≤360 msec and/or ≥450 msec measured at screening or day -2.
2. Exclusion criteria related to cardiac function include the following:

   * The subject has a known clinically significant (in the opinion of the investigator) cardiovascular disorder, including coronary artery disease, valvular heart disease, cardiomyopathies, or an ECG abnormality suggestive of prior myocardial infarction, angina pectoris, chamber enlargement, or hypertrophy. Notwithstanding, subjects with known significant disorders will be excluded.
   * The subject has a known clinically significant arrhythmia or rhythm disturbance observed on the screening and/or day -2 12-lead ECG.
   * The subject has a supine pulse rate outside of the range of 40 to 100 bpm (following at least a 10-minute rest) measured at screening or day -2.
   * The subject has a supine blood pressure outside of the range of 90 to 139 mm Hg systolic or 50 to 89 mm Hg diastolic (following at least a 10-minute rest) measured at screening and on day -2. Note: The blood pressure measurement may be repeated up to 3 times to meet eligibility requirements. In this case, the average of these 3 measurements must meet eligibility criteria.
   * The subject reports a history of, or risk factors for, Torsades de Pointes (eg, congestive heart failure, serum electrolyte abnormalities) including a family history of arrhythmia, sudden unexplained death at a young age (before 40 years) in a first-degree relative, or long QT syndrome, or a personal history of syncope.
3. The subject has low serum potassium and/or magnesium and/or corrected calcium blood levels (less than 3.5 milliequivalent/liter (mEq/L), 1.8 mEq/L, and 8.9 mg/dL, respectively) at screening and/or day-2.
4. The subject has any condition that may possibly interfere with drug absorption, distribution, metabolism, or excretion (eg, previous surgery on the gastrointestinal tract [including removal of parts of stomach, bowel, liver, gall bladder, or pancreas] or stomach banding).
5. The subject has an abnormality in medical history, physical examination, biochemistry, hematology, coagulation, serology, or urinalysis at the screening or admission visit that is considered clinically significant by the investigator or meets grades 2-4 Common Terminology Criteria for Adverse Events (CTCAE) v.4 criteria, or in the opinion of the investigator, could interfere with the objective of the study or the safety of the subject. Notwithstanding, the following values must remain within the normal range values (as determined by the Physician Reference Laboratory [PRL]) in order for a subject to be eligible for the study: calcium, magnesium, potassium, creatinine, ALT, AST, GGT, hemoglobin, absolute lymphocyte count, absolute 50 mg/dL in asymptomatic subjects and absolute leukocyte count values as low as 3.1x109/L in African American subjects will be considered for enrollment at the investigator's discretion. Lastly, the upper limit value for exclusion is modified for the following values and is as follows: INR>1.2, total bilirubin>1.2 mg/dL, serum amylase >143 U/L, LDH>261 U/L, and CPK>367 U/L, which do not normalize upon repeat testing, will be exclusionary.
6. The subject has used one of the prohibited drugs, substances or foods as follows:

   * any investigational product within 60 days (or 5 half-lives, whichever is longer) preceding the study
   * any prescription or nonprescription medication (including herbal remedies, vitamins, or dietary supplements) or vaccine within 14 days of the first day of study drug administration (day 1) or within 5 half-lives before the first day of study drug administration, whichever is longer. Exceptions are locally acting medications (eg, topical creams), which are not allowed within 5 days of study drug administration, and the occasional use of acetaminophen (up to 3 g/day) and ibuprofen (up to 1200 mg/day).
   * consumption of grapefruit, grapefruit juice, Seville oranges, pomelo-containing products, within the 14 days prior to day -1 and then throughout the entire study
   * consumption of excessive amounts of alcoholic beverages, defined as more than 3 drinks per day (beer, wine, or distilled spirits), or unwillingness to comply with the restricted use of alcohol during the study (96 hours prior to admission and until 48 hours after the last study drug administration), history of alcoholism, or evidence of drug/chemical abuse
   * positive urine drug (cocaine, amphetamines, barbiturates, opiates, phencyclidine, benzodiazepines, tetrahydrocannabinol), cotinine, or alcohol screen at the screening visit or admission
   * consumption of quinine (eg, tonic water) within 7 days prior to admission
7. The subject has any other condition, which, in the opinion of the investigator, makes the subject inappropriate for the study.
8. Other exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Individually-corrected QT interval (QTcI) | Up to 23.5 hours after the start of study drug infusion on Day 7
  The primary ECG variable and endpoint for this study is the time-matched change from baseline in QTcI method on day 7 at each time point. Holter ECGs will be performed at baseline (day -1) and prior to the start of infusion on day 7 and 1, 2 (end of infusion), 2.5, 3, 4, 5, 6, 8, 12, 16, 20, and 23.5 hours after the start of infusion.

SECONDARY OUTCOMES:
Fridericia-corrected QT interval (QTcF) | Up to 23.5 hours after study drug infusion on Day 7
  QTcF time-matched change from baseline on day 7 at the following time points: 1, 2 (end of infusion), 2.5, 3, 4, 5, 6, 8, 12, 16, 20, and 23.5 hours
Heart rate, PR interval, QRS interval and uncorrected QT interval | Up to 23.5 hours after study drug infusion on Day 7
  Holter ECGs will be performed at baseline (day -1) and prior to the start of infusion on day 7 and 1, 2 (end of infusion), 2.5, 3, 4, 5, 6, 8, 12, 16, 20, and 23.5 hours after the start of infusion.
ECG morphological patterns | Up to 23.5 hours after study drug infusion on Day 7
  Holter ECGs will be performed at baseline (day -1) and prior to the start of infusion on day 7 and 1, 2 (end of infusion), 2.5, 3, 4, 5, 6, 8, 12, 16, 20, and 23.5 hours after the start of infusion.
QTc (QTcI and QTcF) Intervals | Up to 23.5 hours after study drug infusion on Day 7
  The relationship between the placebo-corrected QTc (QTcI and QTcF) change from baseline and plasma concentrations of custirsen (pharmacokinetic/pharmacodynamic analysis). Holter ECGs will be performed at baseline (day -1) and prior to the start of infusion on day 7 and 1, 2 (end of infusion), 2.5, 3, 4, 5, 6, 8, 12, 16, 20, and 23.5 hours after the start of infusion.
Assay sensitivity | Up to 23.5 hours after study drug infusion on Day 7
  A comparison between the active control, moxifloxacin (400 mg), and placebo will also be performed to demonstrate assay sensitivity as required by current regulatory guidance. Holter ECGs will be performed at baseline (day -1) and prior to the start of infusion on day 7 and 1, 2 (end of infusion), 2.5, 3, 4, 5, 6, 8, 12, 16, 20, and 23.5 hours after the start of infusion.
Maximum observed plasma concentration (Cmax) | From Day 1 through the Follow-up Visit (approximately Day 17)
Time to maximum observed plasma concentration (Tmax) | From Day 1 through the Follow-up Visit (approximately Day 17)
Area under the plasma concentration-time curve (AUC0-t) | From Day 1 through the Follow-up Visit (approximately Day 17)
Area under the curve from time 0 to infinity (AUC0-∞) | From Day 1 through the Follow-up Visit (approximately Day 17)
Percentage of AUC0-∞ due to extrapolation from the time of last measurable concentration to infinity | From Day 1 through the Follow-up Visit (approximately Day 17)
Area under the curve from time 0 to 24 hours (AUC0-24) | From Day 1 through the Follow-up Visit (approximately Day 17)
Terminal elimination rate constant (kel) | From Day 1 through the Follow-up Visit (approximately Day 17)
Apparent terminal half life (t½) | From Day 1 through the Follow-up Visit (approximately Day 17)
Apparent volume of distribution (Vz) | From Day 1 through the Follow-up Visit (approximately Day 17)
Apparent total body clearance (CL) | From Day 1 through the Follow-up Visit (approximately Day 17)
Occurrence of Adverse Events | From signing of the informed consent through the Follow-up Visit (approximately 17 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Teva Investigational Site 10565, Lenexa, Kansas, United States